CLINICAL TRIAL: NCT03140293
Title: A Randomized Trial to Determine if Local Anesthesia Decreases Pain Perception in Women Undergoing Chorionic Villus Sampling
Brief Title: Pain Perception During Chorionic Villus Sampling
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Angela Bianco (Other)
Responsible Party: Sponsor-Investigator, Angela Bianco, MD, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-1425
Record Dates: First submitted 2017-03-28; First posted 2017-05-04 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Chorionic Villi Sampling
Keywords: Chorionic villus sampling; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lidocaine Injection (Active Comparator): Injection of lidocaine which is given prior to chorionic villus sampling
  Interventions: Drug: Lidocaine injection
- Gebauer Ethyl Chloride Spray (Experimental): Topical anesthesia will be Gebauer Ethyl Chloride sprayed continuously from 3 - 7 seconds from a distance of 3-9 inches until the skin turns white (not frosting the skin) as per Gebauer package insert instructions.
  Interventions: Drug: Gebauer Ethyl Chloride Spray

INTERVENTIONS:
Drug: Lidocaine injection — Injectable anesthesia is 1-2mL of 2% lidocaine via a 22 gage needle, given at the anticipated site of CVS needle puncture immediately before procedure.
  Arms: Lidocaine Injection
Drug: Gebauer Ethyl Chloride Spray — Gebauer Ethyl Chloride Spray is a topical anesthetic spray which is sprayed continuously for 3-7 seconds from a distance of 3-9 inches at the site where the chorionic villus sampling is expected to take place.
  Arms: Gebauer Ethyl Chloride Spray

SUMMARY:
Chorionic villous sampling is a frequent procedure used for antenatal genetic testing. This procedure is associated with anxiety and fear of pain that can be expected during the procedure, often prejudicing patients against this definitive antenatal testing. It is important to determine if different approaches to pain and anxiety reduction are effective. Currently there is no randomized study to evaluate the efficacy of analgesia for pain reduction during chorionic villous sampling. Multiple studies have been published suggesting that analgesia during the similar procedure of amniocentesis does not significantly reduce pain scores.

DETAILED DESCRIPTION:
Chorionic villous sampling (CVS) is a frequent procedure used for antenatal genetic testing. This procedure is associated with anxiety and fear of pain that can be expected during the procedure, often prejudicing patients against this definitive antenatal testing. It is important to determine if different approaches to pain and anxiety reduction are effective. Previous studies have not shown that local anesthesia affects pain experience during amniocentesis (1-5). There are no randomized studies evaluating interventions for pain reduction during chorionic villous sampling which constitutes an important evidence gap.

The study will be offered to women at <13 weeks gestation, with a singleton fetus who are seen at Mount Sinai Medical Center for chorionic villous sampling. The eligible women will be randomized to one of two groups: use of analgesia using injectable lidocaine or ethyl chloride topical anesthetic spray. This study intends to show that local anesthesia during chorionic villous sampling will not decrease the perception of pain in patients undergoing this procedure.

This trial is trying to determine perception of pain based on use of injectable lidocaine or ethyl chloride anesthetic spray; it is noted that the form of anesthesia may be a factor in perception of pain. The investigators do not know if there is a difference in perception for topical or injectable. If the perceived pain is comparable in topical and injectable, this trial could conclude that both are viable options, and while both present minimal risk to patients, topical is less invasive.

ELIGIBILITY:
Inclusion Criteria:

* <13 week gestation
* Singleton gestations undergoing CVS

Exclusion Criteria:

* Multiple gestations
* More than one attempt of needle insertion
* Allergy or hypersensitivity to local anesthesia

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain perception scores VAS () | day 1
  Procedure pain perception score as measured by the visual analog scale. By means of analysis of the receiver operating characteristic curves on a 100mm VAS: no pain 0-2 mm, mild pain 2-17 mm, moderate pain 17-47 mm, severe pain 47-77 mm, very severe pain 77-96 mm, most severe pain imaginable 96-100 mm
Verbal Rating Scale (VRS) | day 1
  Procedure pain perception score as measured by the Verbal Rating Scale. 0=no pain, 1=mild pain, 2=moderate pain, 3=severe pain, 4=very severe pain, 5=most severe pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Rekawek, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai; Angela Bianco, M.D., Study Director — Ichan School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Csaba A, Bush MC, Saphier C. How painful are amniocentesis and chorionic villus sampling? Prenat Diagn. 2006 Jan;26(1):35-8. doi: 10.1002/pd.1323. PMID 16378331
- [Background] Mujezinovic F, Alfirevic Z. Analgesia for amniocentesis or chorionic villus sampling. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD008580. doi: 10.1002/14651858.CD008580.pub2. PMID 22071854
- [Background] Gordon MC, Ventura-Braswell A, Higby K, Ward JA. Does local anesthesia decrease pain perception in women undergoing amniocentesis? Am J Obstet Gynecol. 2007 Jan;196(1):55.e1-4. doi: 10.1016/j.ajog.2006.08.025. PMID 17240233
- [Background] Van Schoubroeck D, Verhaeghe J. Does local anesthesia at mid-trimester amniocentesis decrease pain experience? A randomized trial in 220 patients. Ultrasound Obstet Gynecol. 2000 Nov;16(6):536-8. doi: 10.1046/j.1469-0705.2000.00240.x. PMID 11169347
- [Derived] Rekawek P, Stone JL, Robles B, Connolly KA, Bigelow CA, Tudela F, Bianco AT. Pain perception during transabdominal chorionic villus sampling: a randomized trial comparing topical ethyl chloride anesthetic spray and lidocaine injection. J Matern Fetal Neonatal Med. 2021 Feb;34(3):339-345. doi: 10.1080/14767058.2019.1607288. Epub 2019 Apr 25. PMID 30983457